CLINICAL TRIAL: NCT02905240
Title: A Multicenter, Double-Blind, Randomized, Saline-Controlled Study of a Single, Intra-articular Injection of Autologous Protein Solution in Patients With Knee Osteoarthritis
Brief Title: Saline-Controlled Study of nSTRIDE APS for Knee Osteoarthritis
Acronym: PROGRESS IV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APSS-44-00
Record Dates: First submitted 2016-09-14; First posted 2016-09-19 (Estimated); Results first posted 2023-10-19 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-10

CONDITIONS: Osteoarthritis
Keywords: Autologous Protein Solution; APS; intra-articular injection; osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- nSTRIDE APS (Experimental): Autologous Protein Solution prepared using the nSTRIDE APS Kit
  Interventions: Device: nSTRIDE APS
- Saline (Other): Saline control
  Interventions: Device: Saline

INTERVENTIONS:
Device: nSTRIDE APS — single intra-articular injection
  Other Names: Autologous Protein Solution
  Arms: nSTRIDE APS
Device: Saline — single intra-articular injection
  Arms: Saline

SUMMARY:
A double-blind, multicenter, randomized, controlled trial (RCT) that will evaluate the efficacy of a single dose of Autologous Protein Solution (APS) in patients with Osteoarthritis (OA) of the knee.

DETAILED DESCRIPTION:
A double-blind, multicenter, randomized, saline-controlled trial (RCT) that will evaluate the efficacy of a single dose of Autologous Protein Solution (APS) in patients with symptomatic osteoarthritis (OA) of the knee who have not been able to get satisfactory pain relief with prior treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 21 and ≤ 80 years old at the time of screening
* Willingness and ability to comply with the study procedures and visit schedules and ability to follow oral and written instructions
* A standing radiograph of the knee showing a Kellgren-Lawrence grade of 2 to 4 and an absence of severe osteoarthritis
* Body Mass Index ≤ 40
* A qualifying WOMAC LK 3.1 pain subscale total score
* Has undergone at least one prior conservative osteoarthritis treatment
* Signed an institutional review board approved informed consent

Exclusion Criteria:

* Presence of clinically observed active infection in the index knee
* Presence of symptomatic osteoarthritis in the non-study knee
* Diagnosed with rheumatoid arthritis, Reiter's syndrome, psoriatic arthritis, gout, ankylosing spondylitis, or arthritis secondary to other inflammatory diseases; HIV, viral hepatitis; chondrocalcinosis, Paget's disease, or villonodular synovitis
* Diagnosed with leukemia, known presence of metastatic malignant cells, or ongoing or planned chemotherapeutic treatment
* Untreated symptomatic injury of the index knee
* Presence of surgical hardware or other foreign body intended to treat arthritis or cartilage-related pathology in the index knee
* Previous cartilage repair procedure on the injured cartilage surface of the index knee
* Arthroplasty or open surgery of the index knee within 6 months of screening
* Intra-articular steroid injection in the index knee within 3 months of screening
* Intra-articular hyaluronic acid injection in the index knee within 6 months of screening
* Other intra-articular therapy in the index knee within 6 months prior to screening
* Orally administered systemic steroid use within 2 weeks of screening
* Planned/anticipated surgery of the index knee during the study period
* Skin breakdown at the knee where the injection is planned to take place
* Pregnant or nursing mothers or women planning on getting pregnant during the time they will be participating in the study
* Participated in any investigational drug or device trial within 30 days prior to screening
* Participated in any investigational biologic trial within 60 days prior to screening

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Actual)
Dates: Start 2016-11; Primary Completion 2019-07 (Actual); Study Completion 2020-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederick M Azar, M.D., Principal Investigator — Campbell Clinic
Locations (27):
- United States (27):
  - University of Alabama, Birmingham, Alabama
  - AVANT Research Associates, LLC, Guntersville, Alabama
  - Tucson Orthopaedic Institute, PC, Tucson, Arizona
  - CORE Orthopaedic Medical Center, Encinitas, California
  - University of California at Los Angeles, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Andrews Research and Education Foundation (AREF), Gulf Breeze, Florida
  - Florida Hospital Orthopaedic Institute and Fracture Care Center, Orlando, Florida
  - Comprehensive Clinical Trials, LLC, West Palm Beach, Florida
  - Orthoillinois, Ltd., Rockford, Illinois
  - Orthopedic & Sports Medicine Center, Elkhart, Indiana
  - OrthoIndy, Greenwood, Indiana
  - Kansas University Medical Center Research Institute, Inc., Kansas City, Kansas
  - Brigham and Women's Mass General Health Care Center, Foxborough, Massachusetts
  - Northwell Health - Great Neck, Great Neck, New York
  - Northwell Health - Lenox Hill, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest School of Medicine, Winston-Salem, North Carolina
  - University of Cincinnati College of Medicine, Cincinnati, Ohio
  - Ohio State University, Columbus, Ohio
  - Joint Implant Surgeons, Inc, New Albany, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - The Campbell Foundation, Germantown, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - Texas Center for Joint Replacement, Plano, Texas
  - University of Virginia, Charlottesville, Virginia
  - OrthoVirginia, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] King W, van der Weegen W, Van Drumpt R, Soons H, Toler K, Woodell-May J. White blood cell concentration correlates with increased concentrations of IL-1ra and improvement in WOMAC pain scores in an open-label safety study of autologous protein solution. J Exp Orthop. 2016 Dec;3(1):9. doi: 10.1186/s40634-016-0043-7. Epub 2016 Feb 9. PMID 26915009
- [Background] van Drumpt RA, van der Weegen W, King W, Toler K, Macenski MM. Safety and Treatment Effectiveness of a Single Autologous Protein Solution Injection in Patients with Knee Osteoarthritis. Biores Open Access. 2016 Aug 1;5(1):261-8. doi: 10.1089/biores.2016.0014. eCollection 2016. PMID 27668131

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During the screening process, potential subjects provided informed consent and were then screened for eligibility. Screening consisted of meeting all inclusion and exclusion criteria, including a WOMAC LK 3.1 pain subscale score ≥ 9 and ≤ 19 and by providing objective physiological evidence of OA using the Kellgren-Lawrence scale (assessed from normal radiographs).
Period: Overall Study
Arm/Group | nSTRIDE APS | Saline
Started | 172 | 160
Completed | 154 | 137
Not Completed | 18 | 23

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | nSTRIDE APS | Saline | Total
Number analyzed (Participants) | 172 | 160 | 332
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.5 (10.3) | 58.6 (9.6) | 58.55 (9.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 90 | 170
  Male | 92 | 70 | 162
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African-American | 14 | 13 | 27
  Asian or Pacific Islander | 5 | 1 | 6
  Native American | 1 | 1 | 2
  Not Specified | 1 | 1 | 2
  Other | 5 | 2 | 7
  White (Hispanic) | 21 | 7 | 28
  White (Non-Hispanic) | 125 | 135 | 260
Region of Enrollment [Number; unit: participants]
  United States | 172 | 160 | 332
WOMAC Pain [Mean (Standard Deviation); unit: points] — The WOMAC LK 3.1 questionnaire is a validated tool commonly used for assessing knee pain, stiffness, and function. The WOMAC pain subscale consisted of five questions scored from 0 to 4. The pain score has a range of 0 (no pain) to 20 (maximal pain).
  points | 11.27 (2.23) | 11.37 (2.11) | 11.32 (2.17)

OUTCOME MEASURES:

1. Primary Outcome: Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Likert (LK) 3.1 Pain Subscale Change From Baseline to 12 Months
Description: The primary objective of this study was to determine whether nSTRIDE APS is superior to Saline with respect to the improvement in mean WOMAC Pain score (change from baseline to 12 Months post-injection raw score). The WOMAC pain subscale consisted of five questions scored from 0 to 4. The pain score has a range of 0 (no pain) to 20 (maximal pain).
Time Frame: Baseline and 12 Months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | nSTRIDE APS | Saline
Number analyzed (Participants) | 172 | 160
score on a scale | -5.6 [-6.3 to -4.9] | -5.4 [-6.2 to -4.6]

2. Secondary Outcome: Visual Analog Scale (VAS) Pain Change From Baseline to 12 Months
Description: The Visual Analogue Scale is a common tool for measuring general pain. A 100 mm line is marked from 0 to 10 in 10 mm increments. Knee pain severity is indicated by drawing a vertical mark at the point on the line that best represents the severity of pain. No pain is indicated by the 0 at the far left, and the worst possible pain is indicated by the 100 at the far right.
Time Frame: Baseline and 12 Months
Population: Number of subjects with a completed VAS pain score at Baseline and at 12 Months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | nSTRIDE APS | Saline
Number analyzed (Participants) | 149 | 134
score on a scale | -25.8 (27.09) | -23.4 (29.14)

3. Secondary Outcome: Outcome Measures in Rheumatology - Osteoarthritis Research Society International (OMERACT-OARSI) Responders
Description: The OMERACT-OARSI Responder Criteria were applied to both treatment groups, categorizing each patient into one of two categories: responder and non-responder. Responders were defined as subjects who achieved a high degree of improvement in pain or in function (improvement of ≥50% and absolute change ≥20), or a moderate degree of improvement in 2 of the 3 response domains (pain, function, global assessment).
Time Frame: 12 months
Population: Number of subjects with complete data at 12 Months to calculate responder status
Measure: Count of Participants; unit: Participants
Arm/Group | nSTRIDE APS | Saline
Number analyzed (Participants) | 149 | 134
Participants
  Responder | 101 | 92
  Non-Responder | 48 | 42

4. Secondary Outcome: Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) LK 3.1 Stiffness Subscale Change From Baseline to 12 Months
Description: The WOMAC stiffness subscale consisted of two questions scored from 0 to 4. The stiffness score has a range of 0 (no stiffness) to 8 (maximal stiffness).
Time Frame: Baseline and 12 Months
Population: Number of subjects with a completed WOMAC stiffness score at Baseline and at 12 Months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | nSTRIDE APS | Saline
Number analyzed (Participants) | 149 | 134
score on a scale | -2.1 [-2.4 to -1.8] | -2.2 [-2.6 to -1.9]

5. Secondary Outcome: EQ-5D Change From Baseline to 12 Months
Description: The EQ-5D is a validated instrument that assesses an individual's current health status and heath related quality of life. The EQ-5D-3L descriptive component assesses five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression over three levels of severity. The EQ visual analogue scale (EQ VAS) assesses the respondent's self-rated overall health state on a scale from 0 (worst imaginable health state) to 100 (best imaginable health state).
Time Frame: Baseline and 12 Months
Population: Number of subjects with a completed EQ-5D score at Baseline and at 12 Months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | nSTRIDE APS | Saline
Number analyzed (Participants) | 149 | 134
score on a scale | 4.62 [2.02 to 7.22] | 4.06 [1.32 to 6.80]

6. Secondary Outcome: Adverse Events
Description: Subjects experiencing at least one AE
Time Frame: 12 months
Population: Intent to Treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | nSTRIDE APS | Saline
Number analyzed (Participants) | 172 | 160
Participants | 94 | 93

7. Post Hoc Outcome: Post-Hoc Pain/Medication Usage Responder Analysis
Description: This criteria is based on the usage of rescue medication and restricted medication/therapy usage and the WOMAC pain subscale percent change from baseline. A patient is considered a non-responder if one or more of the following are true:
  1. Early exit for Knee OA per IDMC determination
  2. WOMAC Pain Percent improvement 27%
  3. Rescue Medication not withheld within 48 hours of the 12 month study visit
  4. Medication/therapy violation at the 12 month visit (New or Continuing)
  5. Rescue medication taken most days or every day, as reported at the 12 month visit
Time Frame: Baseline and 1 Year
Population: Per Protocol population at 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | nSTRIDE APS | Saline
Number analyzed (Participants) | 162 | 151
Participants
  Non-Responder | 65 | 80
  Responder | 97 | 71

ADVERSE EVENTS:
Time Frame: All AEs reported to or identified by investigative center personnel occurring during the study period, beginning on the day of procedure through completion of follow-up, an average of 12 months.
Description: AEs had the onset and resolution date(s) listed (when known), and had their management and outcome documented (where feasible), and were assessed for severity, seriousness, relatedness, and whether they were anticipated. Narratives of SAEs were adjudicated by a Medical Monitor. An Independent Data Monitoring Committee (IDMC) also met periodically to review aggregate and individual subject data related to safety, data integrity and overall conduct of the trial.
Arm/Group | nSTRIDE APS | Saline
All-Cause Mortality (participants affected / at risk) | 1/172 | 1/160
Serious Adverse Events (participants affected / at risk) | 8/172 | 8/160
Other Adverse Events (participants affected / at risk) | 0/172 | 0/160
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | nSTRIDE APS (N=172) | Saline (N=160)
Heart Attack (Cardiac disorders) | 1 (1) | 0 (0) — Cardiac Catherization, Stent Placement and Medication
Death (Investigations) | 1 (1) | 1 (1) — Not Noted
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Excessive Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
GERD and Hiatal Hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) — Nissen Fundoplication
Right Knee Patella Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Contralateral Knee Patella Replacement
Perforated Diverticulitis (Gastrointestinal disorders) | 1 (1) | 0 (0) — Bowel Rest and IV Antibiotics
Acute Cholecystitis (Gastrointestinal disorders) | 1 (1) | 0 (0) — Laproscopic Cholecystectomy
Lap Band Slippage and Diverticulitis (Gastrointestinal disorders) | 0 (0) | 1 (1) — Laparoscopic Revision of Gastric Band
Confusion, Memory Loss (Psychiatric disorders) | 0 (0) | 1 (1)
Respiratory Syncytial Virus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Oral and IV Corticosteroids
Abnormal Cardiac Stress Test (Cardiac disorders) | 0 (0) | 1 (1) — Heart Catheterization
Kidney Stones (Hepatobiliary disorders) | 1 (1) | 0 (0) — Lithotripsy and Medication
Thyroid Mass (Endocrine disorders) | 1 (1) | 0 (0) — Partial Thyroidectomy
Severe Dizziness (General disorders) | 1 (1) | 0 (0) — Gait and Balance training
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0) — Cardio Conversion

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-08-06): https://cdn.clinicaltrials.gov/large-docs/40/NCT02905240/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-06): https://cdn.clinicaltrials.gov/large-docs/40/NCT02905240/SAP_001.pdf